CLINICAL TRIAL: NCT02286466
Title: Mobile Application of Cognitive-Behavioral Therapy (CBT) for Anxiety and Cancer
Brief Title: Mobile App of CBT for Anxiety and Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Clinical Assistant in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-533
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Cancer; Anxiety
MeSH Terms: conditions — Neoplasms; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education Program (Active Comparator): The presence and usage of Health Education Program.
  Interventions: Behavioral: Health Education Program
- CBT Mobile Application (Experimental): The presence and usage of a CBT Mobile Application.
  Interventions: Behavioral: CBT Mobile Application

INTERVENTIONS:
Behavioral: Health Education Program — Participants in the control group will receive a health education program using a tablet computer identical to the intervention group. The content of this program is adapted from a health education intervention used as the control condition for a cognitive behavioral stress and affect management intervention in a NIH-funded randomized controlled trial of a quality of life intervention for patients with advanced prostate cancer (R21CA102761, PI: Penedo). The program consists of the same number of sessions as the intervention group and includes general information about health and well-being. Specifically, control participants will learn information about topics such as healthy eating, exercise, memory and cognition, and side effects in the context of a cancer diagnosis and treatment.
  Arms: Health Education Program
Behavioral: CBT Mobile Application — The CBT intervention is brief, consisting of 6 modules lasting approximately 30 minutes each. Sessions focus on skills for relaxation, coping with cancer-related worries, as well as activity planning and pacing. Prior to starting the program, a trained research assistant will meet with participants in a private office setting to orient them to the software and instruct them on the use of the mobile tablet device. Once patients are comfortable with the functions and features of the mobile app, they will be encouraged to self-administer the intervention on their study-issued tablet at home and during their regularly scheduled oncology visits, for example while receiving chemotherapy infusion or waiting for a doctor's appointment or tests.
  Arms: CBT Mobile Application

SUMMARY:
The proposed study seeks to implement a randomized controlled trial to evaluate the effectiveness and generalizability of an efficacious cognitive-behavioral therapy (CBT) intervention for use as a self-administered mobile application (mobile app) to treat anxiety in patients with metastatic cancer.

DETAILED DESCRIPTION:
Background: Patients with advanced cancer often experience marked anxiety symptoms that are associated with poor quality of life, high physical symptom burden, and complications with medical treatment. We have demonstrated in prior NCI-funded research that individual cognitive-behavioral therapy (CBT), delivered in-person at a tertiary cancer center, is efficacious for treating heightened anxiety in this population. In our randomized-controlled trial of 40 patients with incurable solid tumors, we observed significant reductions in anxiety symptoms per self-report and blind clinician evaluation, with a large effect size underscoring the clinical benefit of the CBT intervention (Cohen's d=0.80). However, timely access to CBT, especially for patients in community clinic settings, is severely limited by shortened life expectancy, scheduling challenges associated with poor functional status, and the lack of trained clinicians and onsite mental health services.

Objective/Hypothesis: The goals of this study are to assess the feasibility and efficacy of delivering CBT for anxiety via mobile application (app) tailored to patients with advanced cancer. We will administer the intervention at two cancer centers, hypothesizing that patients with advanced cancer who receive CBT via mobile app will report significantly greater reductions in anxiety compared to those assigned to a time-matched control group using an online health educational program.

Specific Aims: The primary aims for the proposed project are 1) to adapt our successful CBT intervention for use as a self-administered, mobile application to treat anxiety in patients with advanced cancer; and, 2) to demonstrate the feasibility, efficacy, and generalizability of the CBT mobile app intervention for anxiety compared to an online health education program across two cancer centers (one academic and one community).

Study Design: We will employ sequential mixed qualitative and quantitative methods for intervention adaptation and testing. Specifically, we will dedicate year one of the award to creating and scripting the CBT mobile app intervention for anxiety, which will include multiple electronic features that enhance specificity to patients' individual cancer-related concerns. Up to six patients with metastatic cancer will participate in an initial open pilot study to explore the usability and acceptability of the prototype application. Data from qualitative interviews with these participants will be used to refine and adapt the intervention further. In year two, we will enroll and randomly assign patients with anxiety and metastatic cancer to receive either the CBT mobile app intervention or an online health education program. Patients will self-administer the intervention protocol using a tablet. The target enrollment for the randomized-controlled trial is 120 patients (CBT Mobile App N=60; Control N=60). Randomization will be stratified by study site and disease severity to demonstrate the generalizability of the intervention among patients with diverse malignancies in both academic and community cancer care settings.

Cancer Relevance: According to the American College of Surgeons Commission on Cancer Report (2011), an essential criterion for accreditation as a cancer center is timely patient access to screening and referral for treatment of psychological distress. Yet, most academic and community cancer clinics lack appropriate resources, staff, and training in evidence-based mental health therapies. The proposed project has the potential to address this critical unmet need by adapting an efficacious and clinically-meaningful CBT intervention to a patient-centered and user-friendly platform that can be accessed at home and while patients receive routine oncology care. If successful, our approach could be widely disseminated in a cost-effective manner across multiple oncology settings, greatly improving access to mental health services, especially for patients with cancer in resource-poor communities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a metastatic solid tumor
* Report clinically significant anxiety symptoms (i.e., Hospital Anxiety and Depression Scale (HADS) -Anxiety Subscale > or equal to 8)
* Anxiety is principal psychiatric problem
* At least four weeks after cancer diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Age greater than 18 years
* Ability to read and respond to questions in English

Exclusion Criteria:

* Co-morbid delirium, dementia, or active and untreated major psychiatric condition such as schizophrenia will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Greer, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled at Massachusetts General Hospital Cancer Center in Boston, MA and Lee Memorial Regional Cancer Center in Fort Myers, FL.
Period: Overall Study
Arm/Group | CBT Mobile Application | Health Education Program
Started | 72 | 73
Baseline Clinician Assessment | 72 | 72
Post Self-report | 67 | 68
Completed (Post clinician assessment is collected after completing post self-report survey.) | 65 | 63
Not Completed | 7 | 10
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Declined Clinician Assessment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT Mobile Application | Health Education Program | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.86 (10.08) | 57.03 (12.42) | 56.45 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 17 | 21 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 65 | 68 | 133
  Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 67 | 65 | 132
  Race: African American or Black | 3 | 2 | 5
  Race: Asian | 1 | 3 | 4
  Race: Multiracial | 0 | 1 | 1
  Race: Unknown | 1 | 2 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Grade 0 -- Asymptomatic (Fully active, able to carry on all pre-disease performance without restriction)
  Grade 1 -- Symptomatic but completely ambulatory (Restricted in psychically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work)
  Grade 2 -- Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  Higher score indicates worse performance status.
  Participants
    ECOG = 0 | 26 | 27 | 53
    ECOG = 1 | 39 | 44 | 83
    ECOG = 2 | 7 | 2 | 9
Cancer type [Count of Participants; unit: Participants]
  Gastrointestinal | 23 | 18 | 41
  Gynecologic | 10 | 14 | 24
  Lung | 9 | 15 | 24
  Breast | 8 | 8 | 16
  Melanoma | 10 | 5 | 15
  Sarcoma | 7 | 7 | 14
  Genitourinary | 2 | 5 | 7
  Peritoneal | 3 | 0 | 3
  Thyroid | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Symptoms From Baseline to Post-assessment
Description: Hamilton Anxiety Rating Scale (HAM-A): The HAM-A is a clinician-administered interview used widely in psychiatry research to evaluate anxiety symptoms. Consisting of 14 items that are scored on a scale from 0 (not present) to 4 (very severe), the HAM-A total score ranges from 0 to 56, with higher scores indicating worse anxiety symptoms.
Time Frame: 1) Baseline (within 2 weeks after enrollment), 2) Post-Assessment (8-12 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the Hamilton Anxiety Rating Scale (HAM-A).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CBT Mobile Application | Health Education Program
Number analyzed (Participants) | 65 | 63
Units on a scale | -2.99 (0.96) | -1.85 (0.98)
Statistical Analysis 1: Comparison: CBT Mobile Application vs Health Education Program; Analysis comparing the change in anxiety symptoms (HAM-A) from baseline to post-assessment between groups adjusting for baseline values of criterion outcome and psychotropic medication use; Test type: Superiority; p = 0.412, ANCOVA — a priori threshold p<0.05; Adjusted for baseline values of criterion outcomes and psychotropic medication use; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-1.60 to 3.87], Standard Error of Mean 1.38

2. Secondary Outcome: Change in Quality of Life From Baseline to Post-assessment
Description: Functional Assessment of Cancer Therapy-General: The FACT-G is a valid and reliable self-report, 27-item instrument, consisting of 4 subscales that evaluate physical, functional, emotional and social wellbeing during the past 7 days. Items are scored using a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). The overall score is the sum of the four subscale scores (range 0-108). Higher scores indicate better quality of life, while lower scores indicate worse quality of life.
Time Frame: 1) Baseline (within 2 weeks after enrollment), 2) Post-Assessment (8-12 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the Functional Assessment of Cancer Therapy-General (FACT-G).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CBT Mobile Application | Health Education Program
Number analyzed (Participants) | 67 | 66
Units on a scale | 7.88 (1.76) | 7.87 (1.77)
Statistical Analysis 1: Comparison: CBT Mobile Application vs Health Education Program; Analysis comparing the change in quality of life (FACT-G) from baseline to post-assessment between groups adjusting for baseline values of criterion outcome and psychotropic medication use; Test type: Superiority; p = 0.997, ANCOVA — a priori threshold p<0.05; Adjusted for baseline values of criterion outcome and psychotropic medication use; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-4.99 to 4.96], Standard Error of Mean 2.51

3. Secondary Outcome: Change in Mood Symptoms From Baseline to Post-assessment
Description: Hospital Anxiety & Depression Scale (HADS): The HADS is a self-report instrument that was designed for medical patients and demonstrates adequate psychometric properties for use among individuals with cancer. Comprised of 14-items that are scored on a 4-point Likert scale, the instrument contains two subscales that measure anxiety and depression symptoms in the past week. Total scores for each subscale range from 0 (no distress) to 21 (maximum distress).
Time Frame: 1) Baseline (within 2 weeks after enrollment), 2) and Post-Assessment (8-12 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the Hospital Anxiety & Depression Scale (HADS).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CBT Mobile Application | Health Education Program
Number analyzed (Participants) | 67 | 68
Units on a scale
  HADS-Anxiety Subscale | -4.33 (0.44) | -3.55 (0.44)
  HADS-Depression Subscale | -1.89 (0.39) | -1.41 (0.38)
Statistical Analysis 1: Comparison: CBT Mobile Application vs Health Education Program; Analysis comparing the change in self-report anxiety symptoms on the HADS-Anxiety Subscale from baseline to post-assessment between groups adjusting for baseline values of criterion outcome and psychotropic medication use; Test type: Superiority; p = 0.215, ANCOVA — a priori threshold p<0.05; Adjusted for baseline values of criterion outcome and psychotropic medication use; Mean Difference (Final Values) = 0.78, 95% CI 2-sided [-0.46 to 2.02], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: CBT Mobile Application vs Health Education Program; Analysis comparing the change in self-report depression symptoms on the HADS-Depression Subscale from baseline to post-assessment between groups adjusting for baseline values of criterion outcome and psychotropic medication use; Test type: Superiority; p = 0.379, ANCOVA — a priori threshold p<0.05; Adjusted for baseline values of criterion outcome and psychotropic medication use; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-0.60 to 1.57], Standard Error of Mean 0.55

4. Secondary Outcome: Change in Depression Symptoms From Baseline to Post-assessment
Description: Patient Health Questionnaire-9 (PHQ-9): The PHQ-9 is a brief, validated measure of major depression per the criteria of the Diagnostic and Statistical Manual of Mental Disorders. Patients respond to 9 questions on a scale of 0 (not at all) to 3 (nearly every day). The total scale score ranges from 0 to 27, with higher scores indicating worse depression symptoms.
Time Frame: 1) Baseline (within 2 weeks after enrollment), 2) Post-Assessment (8-12 weeks after baseline)
Population: Analysis population is the number of participants who completed both baseline and post-assessment measures of the Patient Health Questionnaire-9 (PHQ-9).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CBT Mobile Application | Health Education Program
Number analyzed (Participants) | 67 | 68
Units on a scale | -2.29 (0.57) | -2.14 (0.57)
Statistical Analysis 1: Comparison: CBT Mobile Application vs Health Education Program; Analysis comparing the change in depression symptoms on the PHQ-9 from baseline to post-assessment between groups adjusting for baseline values of criterion outcome and psychotropic medication use; Test type: Superiority; p = 0.852, ANCOVA — a priori threshold p<0.05; Adjusted for baseline values of criterion outcome and psychotropic medication use; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-1.45 to 1.75], Standard Error of Mean 0.81

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include event starting on or after Day 0 and on or before Day 90 (3 months).
Arm/Group | CBT Mobile Application | Health Education Program
All-Cause Mortality (participants affected / at risk) | 1/72 | 3/73
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/73
Other Adverse Events (participants affected / at risk) | 0/72 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No